CLINICAL TRIAL: NCT04579835
Title: Twin A Breech External Cephalic Version Intervention Trial
Brief Title: Twin A Breech External Cephalic Version Intervention Trial (TWEXIT)
Acronym: TWEXIT
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Larry Hinkson, Lead Consultant in Obstetrics, Deputy Director, Charite University, Berlin, Germany
Other Study IDs: EA2/116/20
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Breech Presentation; Twin; Complicating Pregnancy
MeSH Terms: conditions — Breech Presentation; Pregnancy Complications | interventions — Version, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: External Cephalic Version — External Cephalic Version Twin A

SUMMARY:
A prospective study assessing the use of external cephalic version for the management of Twin A breech presentation in twin pregnancy.

DETAILED DESCRIPTION:
The primary goal of the study is to determine the success rate of Twin A external Cephalic Version in our obstetric clinic and to determine new favorable sonographic criteria associated with a successful attempt that have not been investigated before.

ELIGIBILITY:
Inclusion Criteria:

* Presence of the written consent of the patients.
* The patients must be over 18 years old .
* No limit in the ability to consent.

Exclusion Criteria:

* Age under 18
* Limited ability to consent
* Placenta previa
* Fetal abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting with Twin A breech presentation to the antenatal clinic
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Success rate of external cephalic version Twin A | 4 hours after external cephalic version
  Mean Percentage (Range 0-100) - Successfully performed external cephalic Versions / Total number of participants

SECONDARY OUTCOMES:
Fetal weight | 30 Minutes before external cephalic version
  Measurement in grams
Fetal Doppler Umbilical Pulsatility Index | 30 Minutes before external cephalic version
  Index mesurent /Ratio
Fetal Doppler Umbilical Resistance Index | 30 Minutes before external cephalic version
  Index mesurent /Ratio
Incidence of pathological cardiotocogramm | 60 Minutes after external cephalic version
  Numerical percentage
Incidence of emergency delivery | 60 Minutes after external cephalic version
  Numerical percentage
Incidence of bleeding | 60 Minutes after external cephalic version
  Numerical percentage
Incidence of contractions | 60 Minutes after external cephalic version
  Numerical percentage
Incidence of rupture of membranes | 60 Minutes after external cephalic version
  Numerical percentage
Pain scores | 60 Minutes after external cephalic version
  Numerical score: Pain scale Linkert score. (0-10 with 10 being extremely painful)
Mode of Delivery | 6 weeks after delivery
  Type of delivery (vaginal or caesarean)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hinkson, FRCOG, Principal Investigator — Charité University Hospital
Locations (1):
- Charité University Hospital, Mitte, Germany

IPD SHARING:
Plan to Share IPD: No